CLINICAL TRIAL: NCT07130357
Title: Prospective Multi-Centre Randomised Controlled Trial on the Effect of Collagen Scaffold Augmentation in Achilles Tendon Rupture Repair
Brief Title: The Effect of Collagen Scaffold Augmentation in Achilles Tendon Rupture Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Dr., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025.416
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles Tendon Rupture; Collagen Scaffold Augmentation; Regeneten; Achilles Tendon Rupture Repair

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will undergo Achilles tendon repair with Collagen Scaffold Augmentation.
  Upon diagnosis of an Achilles tendon rupture, the participant will receive a temporary slab and surgical repair will be scheduled, and the operation will be performed under general anaesthesia with the patient lying prone. The ruptured ends of the right Achilles tendon will be marked, and a 3 cm longitudinal skin incision will be made along the medial border of the tendon. A standardized end-to-end direct surgical repair using non-absorbable sutures in a 2-strand core in a krackow locking fashion will be performed. The bioinductive collagen scaffold will be placed over the repair site and secured with soft tissue anchors. The surgical site will be closed in layers using 3-0 vicryl and 4-0 ethilon.
  The patient will be discharged the following day and will follow a standardized rehabilitation plan by our physiotherapist. The rehabilitation is split into 4 phases: the protect
  Interventions: Device: Collagen Scaffold; Procedure: Achilles tendon repair
- Control Group (Active Comparator): Participants in the control group will undergo Achilles tendon repair using the same method as the intervention group, only without the additional collagen scaffold augmentation. The rehabilitation protocol will also be identical to the intervention group.
  Interventions: Procedure: Achilles tendon repair

INTERVENTIONS:
Device: Collagen Scaffold — The bioinductive collagen scaffold will be placed over the repair site and secured with soft tissue anchors.
  Arms: Intervention group
Procedure: Achilles tendon repair — Upon diagnosis of an Achilles tendon rupture, the participant will receive a temporary slab and surgical repair will be scheduled, and the operation will be performed under general anaesthesia with the patient lying prone. The ruptured ends of the right Achilles tendon will be marked, and a 3 cm longitudinal skin incision will be made along the medial border of the tendon. A standardized end-to-end direct surgical repair using non-absorbable sutures in a 2-strand core in a krackow locking fashion will be performed. The surgical site will be closed in layers using 3-0 vicryl and 4-0 ethilon.

SUMMARY:
This prospective multicenter randomized controlled trial evaluates the clinical efficacy of collagen scaffold augmentation in surgical repair for acute Achilles tendon ruptures. The study will enroll 48 adult participants randomly assigned to either the intervention group (surgical repair with collagen scaffold augmentation) or the control group (standard surgical repair without scaffold). The primary outcome is tendon function assessed using the VISA-A score, while secondary outcomes include tendon healing characteristics measured by ultrasound (thickness, neovascularity), calf muscle strength, ankle range of motion, and complication rates. Follow-up assessments will be conducted at 6 weeks, 3 months, 6 months, and 12 months post-surgery. The study aims to determine whether collagen scaffold augmentation enhances tendon healing and functional recovery compared to conventional repair methods, potentially offering a improved treatment approach for Achilles tendon injuries.

DETAILED DESCRIPTION:
This study is a prospective multi-center randomized controlled trial investigating the effects of collagen scaffold augmentation in surgical repair of acute Achilles tendon ruptures. The research builds upon existing clinical experience and literature suggesting that while surgical techniques have improved mechanical stability of repaired tendons, biological healing remains a limiting factor in recovery. The trial will compare two treatment approaches: one group will receive standard surgical repair augmented with a collagen scaffold, while the control group will undergo conventional repair without scaffold augmentation.

A total of 48 participants will be recruited from five hospitals and randomly assigned to either group with a 1:1 allocation ratio. The surgical procedure involves end-to-end tendon repair using non-absorbable sutures, with the intervention group additionally receiving a bioinductive collagen scaffold placed over the repair site. All participants will follow the same standardized rehabilitation protocol divided into four phases: protection, early loading, strengthening, and return to function.

Intervention Group:

Participants in the intervention group will undergo Achilles tendon repair with Collagen Scaffold Augmentation.

Upon diagnosis of an Achilles tendon rupture, the participant will receive a temporary slab and surgical repair will be scheduled, and the operation will be performed under general anaesthesia with the patient lying prone. The ruptured ends of the right Achilles tendon will be marked, and a 3 cm longitudinal skin incision will be made along the medial border of the tendon. A standardized end-to-end direct surgical repair using non-absorbable sutures in a 2-strand core in a krackow locking fashion will be performed. The bioinductive collagen scaffold will be placed over the repair site and secured with soft tissue anchors. The surgical site will be closed in layers using 3-0 vicryl and 4-0 ethilon.

The patient will be discharged the following day and will follow a standardized rehabilitation plan by our physiotherapist. The rehabilitation is split into 4 phases: the protection phase, early loading phase, strengthening phase and return to function phase. This plan includes non-weight-bearing walking for 2 weeks, partial weight-bearing walking for 4 weeks, then full weight-bearing walking.

Control Group:

Participants in the control group will undergo Achilles tendon repair using the same method as the intervention group, only without the additional collagen scaffold augmentation. The rehabilitation protocol will also be identical to the intervention group.

The primary outcome measure is the Victorian Institute of Sports Assessment-Achilles (VISA-A) score, which evaluates pain, function, and sporting activity. Secondary outcomes include surgical complications, Foot and Ankle Outcome Score (FAOS), ultrasound measurements of tendon thickness and neovascularity, shear wave elastography for tendon elasticity, Achilles tendon resting angle, calf muscle strength, ankle range of motion, and photoacoustic imaging of tendon oxygen saturation. Participants will be assessed at baseline, 6 weeks, 3 months, 6 months, and 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Achilles tendon rupture.
2. Age > 18 and able to provide written informed consent.

Exclusion Criteria:

1. Hypersensitive to bovine-derived materials.
2. Prior foot/ankle surgery or intervention within 1 year
3. Ongoing litigation regarding current injury
4. Active psychological or physical condition pre-empting participation, including psychosis, mental retardation, stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment (VISA-A) | 6 weeks and 3, 6, 12 months after surgery
  The primary outcome is the score of the Victorian Institute of Sports Assessment - Achilles (VISA-A) questionnaire, which is explicitly designed for Achilles tendon. VISA-A will be used to evaluate pain and symptom severity with activity in participants with Achilles tendon rupture. Chinese-speaking participants will complete the validated Chinese VISA-A questionnaire . The VISA-A questionnaire covers three domains associated with AT: pain, function, and sporting activities. A deterioration in self-reported pain, function and sporting activities is the critical reason patients with Achilles tendon rupture come for medical consultation. Improving questions covered in VISA-A is often the rehabilitation goal for these patients.

SECONDARY OUTCOMES:
Surgical complications | During surgery
  Surgical complications will be recorded, such as would problems and early re-ruptures. Based on current evidence, approximately 1 in 9 patients undergoing operative repair of an acute Achilles tendon rupture developed a postoperative complication.
Foot and Ankle outcome scores (FAOS) | 6 weeks and 3, 6, 12 months
  The Foot and Ankle Outcome Score (FAOS) is a open-source, validated piece of instrument to evaluate overall foot and ankle function . It is extensively used in foot and ankle clinical research and is calculated using multiple Likert scale questions which are organized into 5 sub-categories: symptoms, pain, activities of daily living (ADL), sports and quality of life (QOL). The answers in each subcategory are then converted into a score from 0 to 100; with 100 resembling no symptoms and 0 resembling severe symptoms.
Ultrasound measure of tendon thickness | 6 weeks and 3, 6. 12 months
  B-mode ultrasound will be used to locate and measure the maximum thickness of the Achilles tendon (4-9mm) using a greyscale sonographic image. To minimize anisotropic effect, the transducer will be adjusted to ensure the ultrasound beam is perpendicular to the tendon fibers.
Ultrasound measurement of tendon neovascularity | 6 weeks and 3, 6 ,12 months
  Doppler mode is used to measure tendon neovascularity. The transducer is placed perpendicular to obtain a sagittal view of the Achilles tendon. The assessor screens the tendon for the area of maximum Doppler flow and takes a sonographic image. The Öhberg score is then determined during the US examination. Scores range from 0 to 3, with a higher score indicating more Doppler flow in the peritendinous and intratendinous tissues. Pressure from the transducer will be kept to a minimum to prevent occlusion of neovascularization
Ultrasound measurement of tendon elasticity | 6 weeks and 3, 6, 12 months
  Shear wave elastography (SWE) is a technique used to quantify the stiffness of soft tissue and provide objective, quantitative data for clinical references. It works by using a focused ultrasound beam to generate shear waves within the tissues, and measuring the velocity of their propagation. To measure the stiffness of a tendon, the optimal scan plane must first be identified, and the SWE function is then activated with a measurable range of stiffness standardized at 0-600 kPa. An electrogram is obtained and stored, and the stiffness of the tendon is measured using a Q-box tool. The Q-box is circular and set to 2 mm in diameter, covering only the Achilles tendon without including adjacent soft tissues. The mean stiffness of the tendon is measured for each Q-box.
Achilles tendon resting angle | 6 weeks and 3, 6, 12 months
  Achilles tendon resting angle will be measured in flexed positions . The participant will be positioned prone with the knee passively flexed to 90 degrees on visual inspection. A goniometer will be placed on the lateral, plantar aspect of the foot is used to measure the foot angle. The stationary arm of the goniometer is aligned with the lateral midline of the lower leg, extending towards the knee, while the movable arm is aligned with the calcaneal tuberosity, parallel to the long axis of the foot. To ensure accuracy, the measurement is repeated two to three times, and the average resting angle is calculated.
Calf muscle strength | 6 weeks and 3, 6, 12 months
  Two tests will measure calf muscle strength. At weeks 6 and 3, and 6 months and 1 year, a handheld dynamometer will measure strength while lying down. At 6- and 12-month follow-up, a heel raise test will measure strength. Participants will raise their heels until they tire, with two fingertips per hand on a wall for balance. The heel raise will be done at a rate of 30 per minute, 2 seconds each, and following a metronome
Ankle range of motion | 6 weeks; 3, 6, 12 months
  The weight-bearing lunge test measures ankle dorsiflexion ROM and gauges the flexibility of the gastrocnemius and soleus muscle complex. It is a standardised test that involves standing with heels on the ground and knees aligned with the second and great toe. Participants lunge forward until their knee makes contact with the wall without lifting their heel. The distance between the big toe and the wall is then measured using a ruler
Jump test | 6 weeks; 3, 6, 12 months
  Participants will perform three one-legged counter-movement jumps on a pressure mat (Tekscan, USA) with jump height (cm) calculated from flight time. After demonstration and submaximal practice jumps, the patient executed maximal jumps from a standing position by rapidly squatting (flexing knee/hip/ankle) before exploding upward. The highest jump was recorded, with NPRS-reported Achilles tendon pain immediately post-test.
Tendon oxygenation and vascularity | 6 weeks; 3, 6, 12 months
  The pathological tendon's oxygenation and vascularity were quantified using a multiwavelength photoacoustic ultrasound (PAUS) system equipped with a 7Hz probe and dual-wavelength LED sources (850nm/750nm). The participant assumes a prone position with heels extended beyond the examination table. The probe is positioned on the target tendon, with mode-specific presets selected ("Deep PA" for vascularity at 850nm; "Deep Oxy" for oxygenation at 750nm). Each 20-second acquisition captures 200 frames, with two repeated scans per mode to ensure data reliability.
Thermographic tendon temperature | 6 weeks; 3, 6, 12 months
  Participants will be advised to avoid physical exercise and hot baths before the procedure to ensure data reliability. Each participant will rest in a seated position for 10 minutes followed by 2 minutes without socks. The room will be maintained at 20-24°C. The infrared camera will be positioned one meter from the participant, using a ThermaCam FLIR-T8210. Images will be analyzed with ThermaCAM Researcher Pro 2.8 SR-1 software, and a rectangular area covering the Achilles tendon will be used for temperature assessment.
Achilles Tendon Total Rupture Score | 6 weeks; 3, 6, 12 months
  The Achilles Tendon Total Rupture Score (ATRS) is a validated patient-reported outcome measure specifically designed to assess functional recovery in patients with complete Achilles tendon ruptures. This 10-item questionnaire evaluates symptoms and physical activity limitations, with each item scored on a 0-10 Likert scale (0 = severe disability/unable to perform, 10 = no disability/full function), yielding a total score ranging from 0 (worst) to 100 (best). The ATRS covers three key domains: pain (during rest and activity), functional impairment (walking, stair climbing, running, jumping), and patient confidence in the affected limb.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol